CLINICAL TRIAL: NCT03947528
Title: A Single-dose, Comparative Bioavailability Study of Two Formulations of Sarpogrelate HCl 300mg Tablets Under Fed Conditions
Brief Title: Bioavailability Study of Two Formulations of Sarpogrelate HCl 300mg Tablets Under Fed Conditions
Acronym: Sarpogrelate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DDS18-039BE
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anpl-one SR Tab. 300mg (Experimental): a single oral dose administration in healthy volunteers under fed condition
  Interventions: Drug: Sarpogrelate HCL 300mg
- Sarpodipil SR Tab. 300mg (Active Comparator): a single oral dose administration in healthy volunteers under fed condition
  Interventions: Drug: Sarpogrelate HCL 300mg

INTERVENTIONS:
Drug: Sarpogrelate HCL 300mg — a single oral dose administration in healthy volunteers under fed condition

SUMMARY:
A Single-dose, Comparative Bioavailability Study of Two Formulations of Sarpogrelate HCl 300mg Tablets Under Fed Conditions

DETAILED DESCRIPTION:
To evaluate the bioequivalence of two formulations of Sarpogrelate HCl 300mg after a single oral dose administration in healthy volunteers under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, male and female subjects, 19 years of age or older
* BMI ≥ 18.0 and ≤ 30.0 kg/m2.
* Females who participate in this study will be of childbearing or non- childbearing potential

Exclusion Criteria:

* Know history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the investigator, would jeopardized the safety of the subject or impact the validity of the study results

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-05-13 (Estimated); Study Completion 2019-05-13 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration | 0~24hours
  Maximum Plasma Concentration
Area under the plasma concentration versus time curve | 0~24hours
  Area under the plasma concentration versus time curve

CONTACTS AND LOCATIONS:
Locations (1):
- Daewoong pharmatceutical, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No